CLINICAL TRIAL: NCT02033941
Title: Phase II Grape Seed Extract as Anti-Oligomerization Agent in Alzheimer's Disease
Brief Title: Phase 2 Study to Examine Grape Seed Extract as an Anti-Oligomerization Agent in Alzheimer's Disease (AD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulty with enrollment due to pandemic.
Sponsor: Hillel Grossman (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Hillel Grossman, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 09-0307; 5R21AT005510 (NIH)
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Grapeseed Extract; Clinical Trial; Meganatural-AZ; anti-oligomerization; Phase 2; Dietary Supplement; Nutraceutical
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Meganatural-Az Grapeseed Extract (Active Comparator): Meganatural-Az® doses: 30mg / day for 2 weeks; 4 weeks of 600 mg/day, 4 weeks 1000mg / day
  Interventions: Drug: Meganatural-Az Grapeseed Extract
- Placebo (Placebo Comparator): Subjects receive capsules identical in appearance to the active agent with the same incremental schedule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Meganatural-Az Grapeseed Extract — Meganatural-Az® doses: 30mg / day for 2 weeks; 4 weeks of 600 mg/day, 4 weeks 1000mg / day
  Other Names: Grapeseed Polyphenolic Extract; Grapeseed Phenol Extract; GSPE
  Arms: Meganatural-Az Grapeseed Extract
Drug: Placebo — Subjects receive capsules identical in appearance to the active agent with the same incremental schedule
  Arms: Placebo

SUMMARY:
Alzheimer Disease (AD) is a progressive brain disease generally known as senile dementia. Our proposed study will establish safety and pharmacokinetics of Meganatural-AZ GSPE in AD subjects. As secondary measures, we will also provide the essential human data to guide the design of future studies to test the efficacy of GSPE in mitigating cognitive deterioration in AD patients.

DETAILED DESCRIPTION:
This study aims to establish the safety and pharmacokinetics of Meganatural-Az® GSPE in subjects with Alzheimer's disease. As a secondary goal, clinical and biomarker indices of therapeutic efficacy will also be evaluated. The proposed study will provide the essential human data necessary to guide the design of future studies testing the efficacy of GSPE in mitigating cognitive deterioration in AD patients.

ELIGIBILITY:
Inclusion Criteria:

* NINCDS/ADRDA criteria for probable AD
* MMSE between 12-26
* Treatment with a cholinesterase inhibitor or an NMDA (N-methyl-D-asparate) antagonist with stable dose for at least 12 weeks
* Home monitoring available for supervision of medications
* Caregiver available to accompany patient to all visits and willing to participate in study as informant
* Fluent in English or Spanish
* Medical stability for this study as confirmed by review of records, internist's physical exam, neurological exam, and laboratory tests
* Stable doses of non-excluded medication
* No evidence of hepatic insufficiency
* Able to swallow oral medications
* Ability to participate in the informed consent process

Exclusion Criteria:

* History of hypotension or unstable hypertension
* Active hepatic or renal disease
* Use of another investigational drug within the past two months
* History of clinically significant stroke
* History of seizure or head trauma with disturbance of consciousness within the past two years
* Major mental illness including psychotic disorders, bipolar disorder, or major depressive episode that is not in remission for less than 12 months
* Women of child-bearing age unless using effective birth control or at least one year post-menopausal or surgically menopausal
* Any ferrous or metallic materials which are contraindicated for MRI

Medication Exclusions

* Current use of drugs with significant anticholinergic or antihistaminic properties

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic analysis | up to 22 months
  the pharmacokinetics and effects of Meganatural-Az® on tau and abnormally phosphorylated tau CSF concentrations
primary safety evaluations | up to 22 months
  adverse effects reporting

SECONDARY OUTCOMES:
AD Biomarkers | up to 22 months
  β-amyloid (Aβ) in plasma and in cerebral spinal fluid (CSF) specimens
cognitive and functional assessments | up to 22 months
  cognitive and functional assessments including the ADAS-cog, ADCS CGIC, MMSE, and ADL.

CONTACTS AND LOCATIONS:
Overall Officials: Hillel Grossman, MD, Principal Investigator — Mount Sinai School of Medcine; Samuel Gandy, MD/PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Alzheimer's Disease Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No